CLINICAL TRIAL: NCT03050476
Title: Preventing Oxidative Stress-induced Ischemic Injury- and Systemic Inflammation Complications During and After Invasive Cardiac Surgery With Alkaline Phosphatase (APPIRED III)
Brief Title: Preventing Systemic Inflammation After Cardiac Surgery With Alkaline Phosphatase
Acronym: APPIRED-III
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alloksys Life Sciences B.V. (Industry)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NUH-ALS-2015-04
Record Dates: First submitted 2017-01-24; First posted 2017-02-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Systemic Inflammation; Cardiopulmonary-bypass
Keywords: side-effects; heart-lung machine; alkaline phosphatase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESCAP® (Experimental): Bolus of 1000 IU of bovine intestinal alkaline phosphatase on induction of anaesthesia, followed by an infusion with a sum of 10,000 IU/day over the next 24 or 96 hours.
  Interventions: Drug: RESCAP®
- Placebo (Placebo Comparator): Bolus of of media on induction of anaesthesia, followed by an infusion of media over the next 24 or 96 hours.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RESCAP® — intravenous application before, during, and for 24 or 96 hours after heart surgery
  Arms: RESCAP®
Drug: placebo — intravenous application before, during, and for 24 or 96 hours after heart surgery
  Arms: Placebo

SUMMARY:
Study should demonstrate that alkaline phosphatase reduces the incidence and extent of acute kidney injury after cardiopulmonary bypass (CPB) as defined by the AKIN criteria.

DETAILED DESCRIPTION:
After cardiac surgery under cardiopulmonary bypass (CPB) patients often show impairments of the immune system. Compared to placebo, CPB patients given alkaline phosphatase will have reduced composite endpoint of acute kidney injury (AKI), late extubation, gastrointestinal or neurological complications within 7 days and AKI within 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery with planned cardiopulmonary bypass
* Additive Euroscore II ≥ 3 OR at least 3 surgical cardiac interventions are planned
* Ability to provide informed consent (not incapacitated)

Exclusion Criteria:

* Already on renal replacement therapy
* Patients with chronic kidney disease defined as estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m2 [ CKD stage > 3 ]
* Patients who are pregnant or lactating
* Concurrent enrollment in another clinical trial
* Known allergic reaction to bovine alkaline phosphatase or patient is vegetarian or vegan
* Patients with ongoing infections or current use of steroids
* Patients with high-risk emergency surgery or with follow-up procedures already planned at admission (like e.g. TEVAR)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with acute kidney injury | 90 days
  AKIN criteria: Rise in serum creatinine of by 0.3 mg/dl or 26 µmol/L in 48 hours/ a percentage increase in the serum creatinine concentration of more than 50 percent or a drop in urine output to 0.5 ml/kg/hour for 6 hours
reach haemodynamic stability | 7 days
  Demonstrate that RESCAP® intervention reduces the time at ICU to reach haemodynamic stability

SECONDARY OUTCOMES:
cost-related outcome | 30 days
  Cost (SGD) incurred on renal replacement therapy, ICU and hospital stay
levels of a set of inflammatory markers | 4 days
  IL-6, IL-8, IL-10, IL-17, TNF-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Ruud Brands, PhD, Study Chair — Alloksys Life Sciences BV . President; Dominik Wiedemann, Prof.Dr., Principal Investigator — Universitätsklinikum St. Pölten, Austria
Locations (21):
- Dept. Cardiothoracic Surgery , Monash Medical Centre, Clayton, Melbourne, Australia
- Austria (2):
  - Division of Cardiac Surgery, Department of Surgery, LKH Medical University of Graz, Graz
  - MedUniWien / AKH-Wien, Vienna
- Belgium (5):
  - Department of Intensive Care, CHU Saint-Pierre, Université Libre de Bruxelles (ULB), Brussels
  - Department of Intensive Care, Hôpital Universitaire de Bruxelles (HUB), Brussels
  - Hospital ZOL, Genk
  - Dept. of Anesthesia and Intensive Care, AZ Maria Middelares, Ghent
  - Jessa Ziekenhuis,Campus Virga Jesse, Hasselt
- Germany (2):
  - German Heart Centre Munich, Dept.Cardio-Vascular Surgery, Munich, Bavaria
  - Klinik für Herzchirurgie, Universitätsklinik, Leipzig
- Italy (2):
  - U.O.C. Cardiochirurgia e Trapianti di Cuore, Azienda Ospedaliera San Camillo Forlanini, Roma
  - Policlinico Gemelli, Institute Cardiology, Roma
- Institut Jantung Negara (IJN , Natl. Heart Inst.), Kuala Lumpur, Malaysia
- Netherlands (2):
  - Dept. Cardiothoracic Surgery, Maastricht University Medical Centre, Maastricht, Limburg
  - Catharina Ziekenhuis, Cathreine R&D, Heartcentre, Eindhoven
- Hospital de Santa Marta, Lisbon, Portugal
- Russia (3):
  - State Autonomous Healthcare Institution "Interregional Clinical Diagnostic Center", Kazan'
  - Federal State Budgetary Military Educational Institution of the Higher Education, Saint Petersburg
  - Almazov Heart Center, Saint Petersburg
- National University Hospital (NUH),, Singapore, Singapore
- Jefe de Servicio de Cirugía Cardiovascular, Hospital Universitario La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No